CLINICAL TRIAL: NCT03525379
Title: Evaluating the Clinical Efficacy of Resveratrol in Improving Metabolic and Skeletal Muscle Function in Patients With Heart Failure
Acronym: REV-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Diagnostic
Other Study IDs: REV-HF-2015-1
Record Dates: First submitted 2018-02-01; First posted 2018-05-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Congestive Heart Failure Chronic
Keywords: Skeletal Muscle Blood Flow; (calf muscle) targeted exercise
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: After providing written informed consent, patients who qualify will be randomized via the web-based system coordinated by Research Electronic Data Capture (REDCap) at the University of Alberta. A patient's eligibility will be confirmed and a unique identifier will be assigned.
  Blinding of the patients and study personnel is preserved by using matching placebo capsules. Clinical outcomes will be adjudicated by a Clinical Events Committee, and core laboratories will assess the CMR measures and biomarkers independently and blinded to treatment assignment.
Who Masked: Participant, Care Provider
Masking Description: The randomization codes will be maintained in REDCap. The principal investigator will have authority to unblind patients if safety concerns arise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): 1) Resveratrol- (Transmax) trans- resveratrol (Biotivia Longevity Bioceuticals, LLC, New York, USA) in cellulose capsules. One capsule will be taken orally 2 times per day (BID) for 8 weeks.
  Interventions: Drug: Resveratrol; Drug: Placebo
- Placebo (Placebo Comparator): 2) Placebo- 500mg (Biotivia Longevity Bioceuticals, LLC, New York, USA) in cellulose capsules. One capsule will be taken orally 2 times per day (BID) for 8 weeks.
  Interventions: Drug: Resveratrol; Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — Subject participation will be approximately 10 weeks in duration. Participants will be randomized to receive one treatment: either resveratrol for 8 weeks OR placebo for 8 weeks. There will be a 2-week run-in period prior to the treatment period.
  The schedule for the study is:
  Week 0 Screening and randomization Weeks 1-2 Run-in; no treatment Weeks 3-10 Treatment Phase (resveratrol or placebo)
  Other Names: (Transmax) trans- resveratrol
Drug: Placebo — Participants will be randomized to receive one treatment: either resveratrol for 8 weeks OR placebo for 8 weeks. There will be a 2-week run-in period prior to the treatment period.
  Other Names: Subject participation will be approximately 10 weeks in duration. Participants will be randomized to receive one treatment: either resveratrol for 8 weeks OR placebo for 8 weeks

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial evaluating the effect of resveratrol on metabolic and skeletal muscle function. Patients will be randomized and allocated to either resveratrol or placebo, for 8 weeks with a 2-week run-in period before the intervention period (to ensure they are not on any nutritional supplement that contains resveratrol).

DETAILED DESCRIPTION:
Trial Objectives Primary outcome- Change in Isolated Skeletal Muscle Blood Flow, Oxygen Extraction and Consumption and Metabolic Rate of Recovery with Exercise by Cardiac MRI (CMR). In order to evaluate potential changes in skeletal muscle vascular function and oxygen extraction with resveratrol therapy, the investigators will use a lower limb (calf muscle) targeted exercise protocol in conjunction with magnetic resonance imaging (MRI)32. MRI will be used to measure, simultaneously, the peak rate of blood flow in the calf muscle along with the whole calf muscle extraction of oxygen, which together are used to determine oxygen consumption. This method allows the determinants of oxygen consumption (blood flow and oxygen extraction) to be evaluated, which is necessary to understand the mechanisms of therapy action.

Secondary outcomes-

1. Change in Vascular Function by CMR. Measurement of aortic distensibility will be used to assess changes in the compliance of vascular system with therapy. Compliance will be defined as the fractional change in cross-sectional area of the aorta over the cardiac cycle (measured at both ascending and descending locations) divided by the corresponding change in pressure (pulse pressure = systolic blood pressure - diastolic blood pressure, measured with arm cuff at time of aorta imaging).
2. Change in Body Composition by CMR. Assessment of adipose and visceral fat content in abdomen and skeletal muscle will be made using multi-echo DIXON magnetic resonance image acquisition with automated fat/water decomposition using VARPO post-processing.
3. Phosphocreatinine (PCr) uptake/recovery on skeletal muscle by CMR. Skeletal muscle metabolism will be measured on a 3T PRISMA MRI system (Peter S Allen MRI Centre) equipped with a plantar-flexion exercise setup and phosphorous imaging capabilities. Supine subjects will perform exercise (toe-push on one leg) until exhaustion. P NMR spectra will be acquired continuously during exercise to measure PCr utilization, change in muscle pH, and most importantly, the recovery rate following exercise. PCr recovery following exercise is a direct measure of substrate utilization and oxygen supply, which is measured as the rate of PCr replenishment. The rate constant (in seconds) characterizes the exponential recovery of PCr to resting values (providing a quantitative measure of oxidative phosphorylation. Normal values from healthy controls are 30-35 seconds with prior studies of patients with HF show values of 76 seconds. A study of reproducibility showed a coefficient of variability of 4.6% for this rate constant (from repeated studies on separate days).
4. Change in LVEF, LVEDV and longitudinal strain by CMR. CMR remains the most precise measure of cardiac structure and function and allows for very small sample sizes to detect changes in important variables such as left ventricular ejection fraction (LVEF), left ventricular end diastolic volume (LVEDV) and longitudinal strain. Longitudinal strain is complimentary to volume and ejection fraction and is increasingly used to detect subclinical changes in heart function even in cases of preserved ejection fraction, and is predictive of HF outcomes. The investigators have reported a coefficient of variability of 2.6% for measurement of ventricular volumes with MRI, similar or better than previous studies, which would enable the measurement of a change of 5 ml in LVEDV with therapy, for example, with only 10 subjects (α=0.05, power=0.95).
5. Distance walked on 6-minute walk test (6-MWT). The 6-MWT is a validated and reproducible clinical endpoint that has been used to demonstrate differences in early phase work of medications such as ACE inhibitors, cardiac resynchronization therapy, and exercise interventions.
6. Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ has been used for multiple large RCT and is sensitive to change, validated in patients with heart failure and linked to prognosis in the short and long-term. A minimal clinically important difference is 5 points.
7. Change in Functional Assessment of Chronic Illness Therapy (FACIT-F). The FACIT-F was developed as a quality of life tool to evaluate small changes in fatigue for patients undergoing anemia or cancer therapy. There are no other validated tools specific to heart failure that address fatigue, despite the principal importance of this symptom. Therefore, the FACIT-F will be used to measure fatigue.
8. Change in Sleep Quality. The Medical Outcomes Study (MOS) Sleep Scale is a patient-reported, non-disease-specific instrument for evaluating sleep outcomes. The MOS Sleep Scale measures subjective experiences of sleep across several different domains.

ELIGIBILITY:
Inclusion Criteria:

1. Male: Given the nature of the project and the need to have normative data for variables that may vary by sex, male patients only will be included.
2. Age: Patients should be 50 to 75 years of age. Patients who are younger or older may have variations in skeletal muscle or activity levels that would increase the variation in functional testing.
3. Clinically diagnosed heart failure with reduced ejection fraction (HFrEF; left ventricular ejection fraction <45%) or heart failure with preserved ejection fraction (HFpEF; left ventricular ejection fraction >45%) as defined by the Alberta HEART study.

Exclusion Criteria:

1. Unable to undergo CMR imaging.
2. CMR exclusions: renal failure [a glomerular filtration rate <30 mL/min)], implantable cardiac device (ICD or CRT), uncontrolled atrial fibrillation or recurrent ventricular arrhythmias).
3. General medical conditions: uncontrolled thyroid disorders, hepatic failure, or myocardial revascularization procedures [coronary angioplasty and/or surgical revascularization in the previous 3 months], cancer/malignancy, or with moderate-severe dementia).
4. Patients taking any of the following: oral anticoagulants, insulin, dihydropyridine calcium channel blockers, sildenafil or midazolam.
5. Patients with allergies to the study products.
6. Patients with hormonal disorders.
7. Unwilling to stop regular use of natural health products or dietary supplements containing resveratrol for 14 days prior to study entry and for the duration of the study.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male: Given the nature of the project and the need to have normative data for variables that may vary by sex, male patients only will be included.
Enrollment: 13 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Change in Isolated Skeletal Muscle Blood Flow | 10 weeks
  In order to evaluate potential changes in skeletal muscle vascular function and oxygen extraction with resveratrol therapy, the investigators will use a lower limb (calf muscle) targeted exercise protocol in conjunction with magnetic resonance imaging (MRI). MRI will be used to measure, simultaneously, the peak rate of blood flow in the calf muscle along with the whole calf muscle extraction of oxygen, which together is used to determine oxygen consumption. This method allows the determinants of oxygen consumption (blood flow and oxygen extraction) to be evaluated, which is necessary to understand the mechanisms of therapy action.
Change in Oxygen extraction and consumption | 10 weeks
  In order to evaluate potential changes in oxygen extraction with resveratrol therapy, the investigators will use a lower limb (calf muscle) targeted exercise protocol in conjunction with magnetic resonance imaging (MRI). MRI will be used to measure, simultaneously, the peak rate of blood flow in the calf muscle along with the whole calf muscle extraction of oxygen, which together is used to determine oxygen consumption. This method allows the determinants of oxygen consumption (blood flow and oxygen extraction) to be evaluated, which is necessary to understand the mechanisms of therapy action.

SECONDARY OUTCOMES:
Vascular Function by CMR | 10 weeks
  Measurement of aortic distensibility will be used to assess changes in the compliance of vascular system with therapy. Compliance will be defined as the fractional change in cross-sectional area of the aorta over the cardiac cycle (measured at both ascending and descending locations)

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Cardiovascular and Stroke Research Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided